CLINICAL TRIAL: NCT02363660
Title: A Randomized, Parallel Design Study to Compare the Safety and Effectiveness of Gardasil When Delivered Per Standard Practice (Full Dose, Intramuscular (IM) Delivery Using a Needle and Syringe) vs. Full Dose, IM Delivery Via Needle-free Jet Injection or Reduced Dose, Intradermal Delivery Via Needle-free Jet Injection
Brief Title: Gardasil Immunogenicity With Needle-Free Injection
Acronym: GINI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GINI Study
Record Dates: First submitted 2014-10-16; First posted 2015-02-16 (Estimated); Last update posted 2023-02-17 (Actual); Status verified 2021-03

CONDITIONS: HIV
Keywords: HIV-uninfected

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (Experimental): will receive standard dose (0.5mL) delivered by standard intramuscular injection using a needle and syringe.
  Interventions: Biological: GINI
- Arm II (Experimental): will receive standard dose (0.5mL) delivered by intramuscular injection using the Pharmajet needle-free Stratis device.
  Interventions: Biological: GINI
- Arm III (Experimental): will receive a reduced-dose (0.1 mL) delivered by intradermal injection using the PharmaJet needle-free Tropis device
  Interventions: Biological: GINI

INTERVENTIONS:
Biological: GINI

SUMMARY:
1. Compare rates of seroconversion and GMTs generated following a 3-dose series of vaccine in women given low doses of vaccine by the ID route with the NFI (Group III) to those women given standard doses by the IM route with a needle and syringe (Group I) at 1 month, 6 months and 18 months following completion of the vaccination series.
2. Compare rates of seroconversion and GMTs generated following a 3-dose series of vaccine in women given standard doses of vaccine by the IM route with the NFI (Group II) to those women given standard doses by the IM route with a needle and syringe (Group I) at 1 month, 6 months and 18 months following completion of the vaccination series.

DETAILED DESCRIPTION:
Primary hypotheses:

The primary goal of this study is to compare the vaccination groups. Using GMTs to measure immunogenicity of the 3 different vaccination regimens, we will test for non-inferiority between Group I and Group II and between Group I and Group III.

Our hypotheses are:

1. GMTs of antibodies to all 4 HPV types (6, 11, 16 and 18) following a 3-dose series of vaccine in women given low doses of vaccine by the ID route with the NFI (Group III) will be non-inferior to GMTs in women given standard doses by the IM route with a needle and syringe (Group I). Non-inferiority criteria will have been satisfied when the upper 95% confidence limit on the ratio of GMTs (GI/GIII) is less than 1.5 for all HPV types.
2. GMTs of antibodies to all 4 HPV types (6, 11, 16 and 18) following a 3-dose series of vaccine in women given standard doses of vaccine by the IM route with the NFI (Group II) will be non-inferior to GMTs in women given standard doses by the IM route with a needle and syringe (Group I). Non-inferiority criteria will have been satisfied when the upper 95% confidence limit on the ratio of GMTs (GI/GII) is less than 1.5 for all HPV types.
3. The proportions of baseline-naïve vaccinees seroconverting to all 4 HPV types (6, 11, 16 and 18) following a 3-dose series of vaccine in women given low doses of vaccine by the ID route (Group III) and standard doses of vaccine by the IM route (Group II) with the NFI will be non-inferior to the seroconversion rates in women given standard doses by the IM route with a needle and syringe (Group I). Non-inferiority criteria will have been satisfied when the upper 95% confidence limit on the difference in proportions is less than 10% for all HPV types.

ELIGIBILITY:
Inclusion Criteria:

1. Thai national
2. Woman
3. Age 18-26 years
4. Has had no more than 5 lifetime sex partners
5. HIV-uninfected
6. Able to complete all of the protocol visits and has signed the consent form

Exclusion Criteria:

1. Known contraindications to vaccination with Gardasil

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Needle-free jet injection technology | 24 months
  The jet injector is based on simple, robust technology employing a spring and requiring no compressed gas, battery, or electricity to generate a liquid needle. PharmaJet has two product lines; one for intramuscular and subcutaneous (IM/SC) delivery of 0.5 mL and one for ID delivery of 0.1 mL. The IM/SC product, called Stratis, was FDA-cleared in 2011 and has a separate reset station to recharge the injector spring, while the ID product, Tropis, is in late stage product development and has the reset function integrated into the injector. Both products employ disposable, single-use, needle-free syringes and filling adapter components. To date the products have been used for routine vaccine delivery as well as in a number of clinical trials (including Inactivated Poliovirus Vaccine (IPV), HPV, and influenza). PharmaJet is working with vaccine manufacturers to co-develop custom pre-fillable syringes, e.g., a tetravalent Dengue vaccine with Inviragen.6

CONTACTS AND LOCATIONS:
Locations (1):
- The Thai Red Cross AIDS Research Centre, Pathum Wan, Bangkok, Thailand